CLINICAL TRIAL: NCT02469038
Title: Randomized, Controlled Study of Ultrasound-Guided Peripheral Venous Access Using AccuCath Versus Ultrasound-Guided Conventional Intravenous Catheter in the Emergency Department
Brief Title: Ultrasound-Guided Peripheral Venous Access Using AccuCath
Acronym: AccuCath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB15-0548
Record Dates: First submitted 2015-06-08; First posted 2015-06-11 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Intravenous Access

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AccuCath catheter (Experimental): We use the AccuCath catheter with ultrasound guidance for IV access for patients in the experimental group.
  Interventions: Device: AccuCath catheter
- Control (Active Comparator): We will use ultrasound-guided conventional IV for patients in the control group.
  Interventions: Device: Control

INTERVENTIONS:
Device: AccuCath catheter — Ultrasound-guided insertion of an AccuCath catheter during a standard of care procedure.
  Other Names: Group A
  Arms: AccuCath catheter
Device: Control — Ultrasound-guided insertion of a conventional IV catheter during a standard of care procedure.
  Other Names: Group B; conventional IV catheter
  Arms: Control

SUMMARY:
While peripheral venous cannulation is among the most common procedures performed in clinical settings, it is estimated that PIV insertion fails for 6 million patients annually. Failure to establish peripheral venous access in the emergency department is a costly problem, leading to delays in diagnostics and treatment and requiring alternative sites for vascular access. These alternative methods can lead to higher complications rates, decreased patient satisfaction, and increased utilization of nursing and physician time. Complications from PIV failure also pose a significant financial burden to the healthcare system.

Ultrasound guidance has been shown to greatly improve the process of localizing vessels for cannulation. In a healthcare climate that is increasingly focused on outcomes and cost-effectiveness, ultrasound-guided peripheral venous cannulation has become not only a viable but often the preferred method in patients with difficult venous access. Nevertheless, studies to date on ultrasound-guided peripheral venous cannulation have revealed some shortcomings, such as premature failure and low first attempt success rates.

The purpose of our study is to assess whether ultrasound-guided cannulation of a AccuCath catheter, which has a coiled tip guidewire, is superior to ultrasound-guided cannulation of a conventional peripheral IV catheter across clinical outcomes relevant to the emergency department setting.

DETAILED DESCRIPTION:
Peripheral venous cannulation is among the most common procedures performed in clinical settings and is a prerequisite for fluid resuscitation, administration of medications, and diagnostic testing [1,2]. In the United States, approximately 300 million peripheral intravenous catheters (PIV) are inserted annually [1], and more than 25% of all visits to the emergency department require intravenous catheters for parenteral fluid administration [3]. Providers in the emergency department have become adept at establishing peripheral venous access, but it is estimated that PIV insertion fails for 6 million patients annually [1].

Many factors are thought to be associated with difficult venous access, which is typically defined to be at least two failed attempts at establishing intravenous access [3]. Intravenous drug abuse, obesity, multiple hospitalizations, and chronic medical problems including diabetes, sickle cell disease, end-stage renal disease, and cancer are predisposing factors for difficult venous access [2-5]. Prior studies have reported prevalence of difficult venous access ranging from 8% to 23% [2-5]. Failure to establish peripheral venous access in the emergency department is a costly problem, leading to delays in diagnostics and treatment and requiring alternative sites for vascular access such as external jugular, intraosseous, or central venous access [3]. These alternative methods can lead to higher complications rates, decrease patient satisfaction, and increase utilization of nursing and physician time [6]. Central venous catheterization, which is often used when traditional venous cannulation methods fail, has an overall complication rate of 15%, and complications include arterial puncture, pneumothorax, deep vein thrombosis, and infection [7,8]. These complications pose a significant financial burden to the healthcare system, as the cost associated with a single central venous catheter related infection in 2002 was estimated to be $34,508 to $56,000 and the median payout for claims resulting from central venous catheter related injuries was $100,7502.

In the past few decades, ultrasound guidance has greatly improved the process of localizing vessels for cannulation, especially in patients with abnormal vascular anatomy or difficult venous access, thereby providing many benefits over landmark-based techniques. Ultrasound guided venous cannulation dates back to 1984, when Legler and Nugent showed that the single pass success rate for internal jugular (IJ) cannulation could be improved to 77.3% using Doppler ultrasound versus 28.6% for the traditional landmark-based approach [9]. Since the report of real-time ultrasonographic guidance of IJ catheter placement by Yonei et al. in 1986 [10], ultrasound guided central venous cannulation has repeatedly been shown to increase success rates, decrease complication rates, and improve patient satisfaction [1,2,11-15]. Based on the advantages offered by ultrasound guidance, the Agency for Healthcare Research and Quality now recommends real-time ultrasonographic guidance for all central venous access [13,16].

The ultrasound-guided approach was adapted for peripheral venous access in the emergency department by Keyes et al. in an uncontrolled study that demonstrated a 91% success rate for ultrasound-guided cannulation of brachial and basilica veins [17]. A subsequent controlled study validated a higher success rate in the ultrasonographic (97%) versus control (33%) group in patients identified to have difficult PIV access and also showed that the ultrasonographic group required less time to successful cannulation, fewer percutaneous punctures, and resulted in greater patient satisfaction than the traditional landmark-based approach [13]. Furthermore, ultrasound-guidance for peripheral venous cannulation has been shown to prevent the need for central venous catheterization in 85% of patients with difficult venous access [2] and used 40% fewer kits per patient than landmark-guided placement of catheters [11,18]. In a healthcare climate that is increasingly focused on outcomes and cost-effectiveness, ultrasound-guided peripheral venous cannulation has become not only a viable but often the preferred method in patients with difficult venous access.

Nevertheless, studies to date on ultrasound-guided peripheral venous cannulation have revealed some shortcomings. Conventional IV catheters placed under ultrasound guidance have been prone to premature failure with failure rates of 8% [7,17] in the first hours after placement and 47% in the first 24 hours, most commonly due to infiltration [7]. These failure rates are significantly higher compared with 2% at 24 hours and 10% at day 4, which has been reported for standard peripheral IV catheters [7,19]. Moreover, while overall success rates range from 90% to 100% with multiple attempts [2,7,13,20], first attempt success rate has been less impressive, ranging from 46% to 71% [13,20]. Our study will assess whether the AccuCath catheter with its integrated guidewire can address these shortcomings and demonstrate superiority over conventional PIV catheters across clinical outcomes relevant to the emergency department setting.

While catheters with guidewires have long been used when placing central and arterial lines, they have largely been absent from PIV placement. The AccuCath catheter is differentiated from a conventional IV catheter in two principal ways. The catheter material consists of polyether block amide, which is a thermoplastic elastomer with softness and flexibility designed to decrease vessel wall irritation and mechanical phlebitis [21]. In addition, the integrated guidewire facilitates catheter insertion and limits vessel damage [21]. A prospective, randomized, controlled study has shown a first attempt success rate of 89% for a catheter with guidewire versus 47% for conventional IV along with lower complication rates of 8% for the cathether with guidewire and 52% for conventional IVs [21]. This study was performed in an inpatient setting on patients receiving elective, non-emergent PIVs [21].

Our study will be important in determining whether AccuCath's superior first attempt success rate and lower complication rate can be replicated in emergent PIVs in the emergency department setting. These improvements could translate to cost savings from decreased utilization of physician and nursing time, fewer number of PIV catheters used, higher patient satisfaction from fewer percutaneous punctures, and less complications from infiltration and phlebitis.

The objectives of the study are to:

1. In patients who fail traditional non-ultrasound IV catheter placement, compare ultrasound-guided cannulation of AccuCath catheters versus ultrasound-guided cannulation of conventional IV catheters in ED patients across the following clinical parameters: first attempt success rate, procedure time from the point of first percutaneous puncture to successful cannulation, total number of percutaneous punctures required for successful cannulation, and total number of IV catheters required for successful cannulation.
2. Assess patient and provider satisfaction with each catheter system on a 5-point Likert scale.
3. Check for clinical and demographic differences between patient groups that were successfully cannulated on first attempt versus those that required multiple attempts.

We hypothesize that:

1. Ultrasound-guided cannulation of AccuCath IV catheters will demonstrate a higher first attempt success rate, require less procedure time, require fewer percutaneous punctures, and utilize fewer catheters than ultrasound-guided cannulation of conventional IV catheters in ED patients.
2. Patients and providers will be more satisfied with AccuCath IV catheters versus conventional IV catheters in the ED setting.
3. There will be no statistically significant clinical and demographic differences between patient groups that are successfully cannulated on first attempt versus those that required multiple attempts.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with IV access need

Exclusion Criteria:

* Lack of decisional capacity (e.g., intoxication, dementia, delirium, developmental delay), prior venous grafts or surgery at target IV site, not an acceptable candidate for ultrasound-guided PIV per Mitchell ED protocol (i.e. 3 failed attempts by nurses- 2 by primary nurse, 1 by senior nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Suh, MD MBA MSc, Principal Investigator — University of Chicago; Gregg Helland, MD, Principal Investigator — University of Chicago; Thomas Spiegel, MD MBA, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikari S, Blaivas M, Morrison D, Lander L. Comparison of infection rates among ultrasound-guided versus traditionally placed peripheral intravenous lines. J Ultrasound Med. 2010 May;29(5):741-7. doi: 10.7863/jum.2010.29.5.741. PMID 20427786
- [Background] Au AK, Rotte MJ, Grzybowski RJ, Ku BS, Fields JM. Decrease in central venous catheter placement due to use of ultrasound guidance for peripheral intravenous catheters. Am J Emerg Med. 2012 Nov;30(9):1950-4. doi: 10.1016/j.ajem.2012.04.016. Epub 2012 Jul 15. PMID 22795988
- [Background] Fields JM, Piela NE, Au AK, Ku BS. Risk factors associated with difficult venous access in adult ED patients. Am J Emerg Med. 2014 Oct;32(10):1179-82. doi: 10.1016/j.ajem.2014.07.008. Epub 2014 Jul 30. PMID 25171796
- [Background] Elia F, Ferrari G, Molino P, Converso M, De Filippi G, Milan A, Apra F. Standard-length catheters vs long catheters in ultrasound-guided peripheral vein cannulation. Am J Emerg Med. 2012 Jun;30(5):712-6. doi: 10.1016/j.ajem.2011.04.019. Epub 2011 Jun 23. PMID 21703801
- [Background] Lapostolle F, Catineau J, Garrigue B, Monmarteau V, Houssaye T, Vecci I, Treoux V, Hospital B, Crocheton N, Adnet F. Prospective evaluation of peripheral venous access difficulty in emergency care. Intensive Care Med. 2007 Aug;33(8):1452-7. doi: 10.1007/s00134-007-0634-y. Epub 2007 Jun 7. PMID 17554524
- [Background] Mahler SA, Wang H, Lester C, Skinner J, Arnold TC, Conrad SA. Short- vs long-axis approach to ultrasound-guided peripheral intravenous access: a prospective randomized study. Am J Emerg Med. 2011 Nov;29(9):1194-7. doi: 10.1016/j.ajem.2010.07.015. Epub 2010 Oct 15. PMID 20951527
- [Background] Dargin JM, Rebholz CM, Lowenstein RA, Mitchell PM, Feldman JA. Ultrasonography-guided peripheral intravenous catheter survival in ED patients with difficult access. Am J Emerg Med. 2010 Jan;28(1):1-7. doi: 10.1016/j.ajem.2008.09.001. PMID 20006193
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Legler D, Nugent M. Doppler localization of the internal jugular vein facilitates central venous cannulation. Anesthesiology. 1984 May;60(5):481-2. doi: 10.1097/00000542-198405000-00016. No abstract available. PMID 6711857
- [Background] Yonei A, Nonoue T, Sari A. Real-time ultrasonic guidance for percutaneous puncture of the internal jugular vein. Anesthesiology. 1986 Jun;64(6):830-1. doi: 10.1097/00000542-198606000-00033. No abstract available. PMID 3717653
- [Background] Miller AH, Roth BA, Mills TJ, Woody JR, Longmoor CE, Foster B. Ultrasound guidance versus the landmark technique for the placement of central venous catheters in the emergency department. Acad Emerg Med. 2002 Aug;9(8):800-5. doi: 10.1111/j.1553-2712.2002.tb02168.x. PMID 12153885
- [Background] Denys BG, Uretsky BF, Reddy PS. Ultrasound-assisted cannulation of the internal jugular vein. A prospective comparison to the external landmark-guided technique. Circulation. 1993 May;87(5):1557-62. doi: 10.1161/01.cir.87.5.1557. PMID 8491011
- [Background] Costantino TG, Parikh AK, Satz WA, Fojtik JP. Ultrasonography-guided peripheral intravenous access versus traditional approaches in patients with difficult intravenous access. Ann Emerg Med. 2005 Nov;46(5):456-61. doi: 10.1016/j.annemergmed.2004.12.026. PMID 16271677
- [Background] Randolph AG, Cook DJ, Gonzales CA, Pribble CG. Ultrasound guidance for placement of central venous catheters: a meta-analysis of the literature. Crit Care Med. 1996 Dec;24(12):2053-8. doi: 10.1097/00003246-199612000-00020. PMID 8968276
- [Background] Mallory DL, McGee WT, Shawker TH, Brenner M, Bailey KR, Evans RG, Parker MM, Farmer JC, Parillo JE. Ultrasound guidance improves the success rate of internal jugular vein cannulation. A prospective, randomized trial. Chest. 1990 Jul;98(1):157-60. doi: 10.1378/chest.98.1.157. PMID 2193776
- [Background] Rothschild JM. Ultrasound guidance of central vein catheterization: making healthcare safer: a critical analysis of patient safety practices. Agency for Healthcare Research and Quality Publication No. 01-E058. http://www.ahrq.gov/clinic/ptsafety.
- [Background] Keyes LE, Frazee BW, Snoey ER, Simon BC, Christy D. Ultrasound-guided brachial and basilic vein cannulation in emergency department patients with difficult intravenous access. Ann Emerg Med. 1999 Dec;34(6):711-4. doi: 10.1016/s0196-0644(99)70095-8. PMID 10577399
- [Background] Thompson DR, Gualtiere E, Deppe S, et al. Greater success in subclavian vein cannulation using ultrasound for inexperienced operators. Crit Care Med. 1994;22:A189.
- [Background] Catney MR, Hillis S, Wakefield B, Simpson L, Domino L, Keller S, Connelly T, White M, Price D, Wagner K. Relationship between peripheral intravenous catheter Dwell time and the development of phlebitis and infiltration. J Infus Nurs. 2001 Sep-Oct;24(5):332-41. doi: 10.1097/00129804-200109000-00008. PMID 11575049
- [Background] Gregg SC, Murthi SB, Sisley AC, Stein DM, Scalea TM. Ultrasound-guided peripheral intravenous access in the intensive care unit. J Crit Care. 2010 Sep;25(3):514-9. doi: 10.1016/j.jcrc.2009.09.003. Epub 2009 Oct 15. PMID 19836193
- [Background] Idemoto BK, Rowbottom JR, Reynolds JD, Hickman Jr RL. The AccuCath Intravenous Catheter System With Retractable Coiled Tip Guidewire and Conventional Peripheral Intravenous Catheters: A Prospective, Randomized, Controlled Comparison. The Journal of the Association for Vascular Access. 2014;19(2):94-102.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AccuCath Catheter | Control
Started | 26 | 24
Completed | 22 | 19
Not Completed | 4 | 5
Not completed — Physician Decision | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AccuCath Catheter | Control | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 33
  >=65 years | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (19.4) | 51.6 (17.5) | 46.9 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 19 | 41
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate
Description: Rate of success of first attempt for IV access
Time Frame: During length of stay in emergency room up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | AccuCath Catheter | Control
Number analyzed (Participants) | 22 | 19
Participants | 17 | 11

2. Secondary Outcome: IV Procedure Time
Description: Procedure time from the point of first percutaneous puncture to successful cannulation
Time Frame: During length of stay in emergency room up to 24 hours
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | AccuCath Catheter | Control
Number analyzed (Participants) | 10 | 8
seconds | 294.5 (217.6) | 740.3 (1222.6)

3. Other Pre Specified Outcome: Total Number of Percutaneous Punctures
Description: Total number of percutaneous punctures required for successful cannulation
Time Frame: During length of stay in emergency room up to 24 hours
Measure: Mean (Standard Deviation); unit: punctures
Arm/Group | AccuCath Catheter | Control
Number analyzed (Participants) | 22 | 19
punctures | 1.4 (0.9) | 1.7 (0.9)

4. Other Pre Specified Outcome: Total Number of IV Catheters
Description: Total number of IV catheters required for successful cannulation
Time Frame: During length of stay in emergency room up to 24 hours
Measure: Mean (Standard Deviation); unit: total number of catheters
Arm/Group | AccuCath Catheter | Control
Number analyzed (Participants) | 22 | 19
total number of catheters | 1.1 (0.3) | 1.6 (1.0)

5. Other Pre Specified Outcome: Patient Satisfaction Data
Description: Patient satisfaction data with each catheter system on a 5-point Likert scale minimum value=1, maximum value=5, higher scores are a better outcome
Time Frame: During length of stay in emergency room up to 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AccuCath Catheter | Control
Number analyzed (Participants) | 22 | 19
units on a scale | 4.2 (1.2) | 3.7 (1.3)

6. Other Pre Specified Outcome: Provider Satisfaction Data
Description: Provider satisfaction data with each catheter system on a 5-point Likert scale minimum value=1, maximum value=5, higher scores are a better outcome
Time Frame: During length of stay in emergency room up to 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AccuCath Catheter | Control
Number analyzed (Participants) | 22 | 19
score on a scale | 4.1 (1.1) | 3.8 (1.2)

7. Other Pre Specified Outcome: Clinical and Demographic Information
Description: medical history
Time Frame: During length of stay in emergency room up to 24 hours
Measure: Number; unit: participants
Arm/Group | AccuCath Catheter | Control
Number analyzed (Participants) | 22 | 19
participants
  Type 1 Diabetes | 0 | 2
  Type 2 Diabetes | 4 | 9
  COPD | 1 | 2
  Smoker | 2 | 3
  Dialysis | 4 | 3
  History of Difficult Needle Stick | 10 | 12
  Hypertension | 5 | 16
  Sickle Cell Disease | 7 | 2
  Congestive Heart Failure | 3 | 5

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | AccuCath Catheter | Control
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/19
Other Adverse Events (participants affected / at risk) | 0/22 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT02469038/Prot_SAP_000.pdf